CLINICAL TRIAL: NCT00417430
Title: Phase II Study of Efficacy of ICI 182,780 (Faslodex) in the Treatment of Systemic Lupus Erythematosus: Clinical, Serologic, Molecular
Brief Title: Efficacy of Faslodex in Treatment of SLE Clinical, Serologic, and Molecular Studies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Center for Rheumatic Disease, Allergy, & Immunology (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Nabih I Abdou, MD, PhD, Center for Rheumatic Disease Allergy & Immunology
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 03-082
Record Dates: First submitted 2006-12-28; First posted 2007-01-01 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Fulvestrant

INTERVENTIONS:
Drug: ICI 182,780 (Faslodex)

SUMMARY:
SLE(Systemic Lupus Erythematosus) is an autoimmune disese that primarily occurs in women(9:1 compared to men). The disease is activated by genetic and environmental factors, yet the female gender is the strongest risk factor. The sex hormone estrogen has been proven in the past to be an enhancer of the immune response. Estrogen serves as a ligand for two specific receptor proteins. Lab studies that we have already done have shown estrogen significantly increases these two ligands in the T cells from SLE females, but not in T cells from normal women. These estrogen-dependent increases are blocked by the estrogen receptor antagonist ICI 182,780. The objective of this research is to investigate if ICI 182,780 alters disease progression and/or activity in females with SLE and may provide a new treatment for women with SLE. This is based on previous work we have done.

DETAILED DESCRIPTION:
This is a double-blind study, involving (goal) 20 women with SLE. All will be premenopausal with regular menstrual cycles. Patients will meet at least four of the criteria of the American Colleges of Rheumatology for classification of SLE. Disease activity will be determined by SLE disease activity index called SLEDAI scores. Patients can take meds to control their disease, but none will be able to take birth control pills/patches, or hormone replacement at the time of the study. The pharmacy will be in control of the blind and 10 will get ICI 182,780 (Faslodex) and 10 will get placebo. Lab will be drawn before each injection and a bone density will be done on injection 1 and 12, the injections will be monthly, depending on the female's cycle. A visit will be done at month 15 to evaluate SLEDAI, and draw lab as well. Each vs will have a SLEDAI done with the clinical evaluation. The injection is 250mg/5cc, which is divided into 2 injections of 2.5cc each, given IM, on day 4-10 of each cycle.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women with SLE
* Without life-threatening manifestations
* With regular menstrual cyles not on hormones of any kind

Exclusion Criteria:

For any of the following:

* Increase of SLEDAI greater than 12
* If life-threatening manifestations occur
* If menstruation ceases

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20
Dates: Start 2004-09; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Improved SLEDAI
Improved Disease Lab parameters
Measurement of the estrogen receptors from start to finish

CONTACTS AND LOCATIONS:
Overall Officials: Nabih Abdou, MD, PhD, Principal Investigator — Center for Rheumatic Disease
Locations (1):
- 4330 Wornall suite 40, Kansas City, Missouri, United States